CLINICAL TRIAL: NCT05911100
Title: Evaluation of the Effectiveness of Medical Rehabilitation of COVID-19 Patients Based on the Study of Individual Physiological Parameters of Oxygen Metabolism and the Reserve Capabilities of the Cardiovascular and Respiratory Systems
Brief Title: State of Oxygen Metabolism, Cardiovascular and Respiratory System Reserve Capacity in Patients Who Underwent COVID-19
Status: Active, not recruiting | Type: Observational
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Other Study IDs: 691-КИ
Record Dates: First submitted 2023-06-18; First posted 2023-06-20 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Covid19; COVID19 Infection
Keywords: covid19; rehabilitation; oxygen metabolism
MeSH Terms: conditions — COVID-19 | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Main: Patients 18 years of age and older who have undergone COVID-19 and who are scheduled for the second stage of rehabilitation at the Federal Research Center for Fundamental and Translational Medicine
  Interventions: Diagnostic Test: Spirography and assessment of pulmonary diffusion capacity; Diagnostic Test: Cardiopulmonary stress test; Diagnostic Test: Computed tomography of the chest organs; Diagnostic Test: Heart echocardiography; Other: SF-36 Quality of Life Questionnaire; Diagnostic Test: Demographic and antropometric measures; Other: Indicators characterizing the severity of the underlying disease

INTERVENTIONS:
Diagnostic Test: Spirography and assessment of pulmonary diffusion capacity — Using the Master Screen Body device you will be asked to take two series of breaths through a special tube for 2-3 minutes. Usually the procedure does not cause any discomfort
Diagnostic Test: Cardiopulmonary stress test — The exercise test is performed on a bicycle ergometer Oxycon Pro. Prior to the test, special sensors for recording the electrocardiogram, a sensor to determine blood saturation, and a cuff to measure blood pressure will be glued on the body. Breathing during the test takes place through a face mask with a built-in gas analyzer sensor. The stress test is conducted up to an individual maximum (according to the age, sex, height and weight of the patient), followed by a recovery period. There is some temporary discomfort associated with performing physical activity. Dyspnea, leg fatigue, and dizziness may occur. Observation continues until full recovery of hemodynamic and gas exchange parameters, in case of appearance of unfavorable symptoms - until their disappearance.
Diagnostic Test: Computed tomography of the chest organs — CT is a method of examination based on X-rays, but unlike conventional X-rays, it gives the most complete picture of the body structure, with less radiation.
  Tomography usually does not cause any unpleasant feelings and is performed in a specialized department.
Diagnostic Test: Heart echocardiography — It's a specific method of ultrasound examination, which consists in examining the heart in real time and usually does not cause any unpleasant feelings
Other: SF-36 Quality of Life Questionnaire — https://clinmedjournals.org/articles/jmdt/jmdt-2-023-figure-1.pdf
Diagnostic Test: Demographic and antropometric measures — Age, sex, height. weight, body mass index (BMI)
Other: Indicators characterizing the severity of the underlying disease — * Severity of underlying disease (mMRC, BODE, SMRT-CO Respiratory Support Need Scale), and comorbidities (cardiovascular disease, diabetes mellitus, chronic obstructive pulmonary disease, chronic kidney disease)
  * Medications taken.

SUMMARY:
This clinical study will create an evidence base for rehabilitation approach, which will be used for restoration of pulmonary ventilation and gas exchange, increase of tolerance to physical load reduced in patients who underwent COVID-19.

The aim of the present clinical study is to evaluate the effectiveness of medical rehabilitation of COVID-19 patients based on the study of individual physiological parameters of oxygen metabolism and reserve capabilities of the cardiovascular and respiratory systems.

DETAILED DESCRIPTION:
After an interview about the possibility of taking part in the study, the patient is presented with an informed consent form, explaining all the questions of interest. In the case of consent to participate in the study, the patient and the researcher fill out all the necessary fields of the two copies of the informed consent and sign it. If necessary, the researcher re-explains any information about the study. One copy of the informed consent remains with the patient, and the second copy is kept by the investigator, as required by Good Clinical Practice.

Once informed consent is obtained, an Individual Registration Card (IRC) is completed for the patient enrolled in the study. Completion of the IRC also continues until completion of the second phase of rehabilitation.

Pulmonary functional tests, cardiopulmonary stress testing (CPT) are performed on day 1 or 2 of inclusion of the patient in the rehabilitation program of "Federal Research Center for Fundamental and Translational Medicine" (FRC FTM) using MasterScreen Pneumo (Jaeger, Germany) and Oxycon Pro ergospirometry systems (Jaeger, Germany), in accordance with international standards. The indexes of external respiration are brought to BTPS conditions, and gas exchange - STPD. The protocol of stress testing is chosen individually, based on the proper values in accordance with the age, sex and anthropometric data of the patient. The study is conducted up to the individual maximum, followed by a recovery period. The anaerobic threshold is determined using the V-slope method. After peak load is reached, it is gradually reduced. Observation is continued until complete recovery of hemodynamic parameters, gas exchange, in case of adverse symptoms - until their disappearance. Repeated testing is performed after the rehabilitation program, before discharge from the FTC MTF.

Thoracic MSCT is performed on day 1-2 of inclusion of a patient into the rehabilitation program of the FRC FTM to assess the lesion of the bronchopulmonary system after COVID-19.

Questionnaires describing the severity of the underlying disease (mMRC respiratory impairment scale, BODE pulmonology risk scale, SMRT-CO respiratory support need scale), and SF-36 quality of life questionnaire are completed at study inclusion and after the rehabilitation program, before discharge from the FRC FTM.

ELIGIBILITY:
Inclusion Criteria:

* pneumonia or acute respiratory distress syndrome caused by SARS-CoV-2
* referral for a second phase of rehabilitation
* signed informed consent of the patient to participate in the study

Exclusion Criteria:

* mental and/or locomotor disorders that make it impossible to adequately perform an exercise test, cooperate with the patient, and interpret the results
* conditions and diseases requiring emergency surgical intervention and/or observation and treatment in the ICU
* patient's refusal to participate in this clinical trial at any stage of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People 18+ years old who have undergone COVID-19 infection and are scheduled for the second stage of rehabilitation at the Federal Research Center for Fundamental and Translational Medicine.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Need for respiratory support according to SMRT-CO criteria. | From enrollment to the end of treatment at 4 to 6 weeks
  The SMART-COP Score for Pneumonia Severity predicts need for intensive respiratory or vasopressor support in community-acquired pneumonia.

SECONDARY OUTCOMES:
Peak oxygen consumption | From enrollment to the end of treatment at 4 to 6 weeks
  Maximum oxygen consumption is the highest amount of oxygen, expressed in milliliters, that a person can consume in 1 minute.
Diffusion capacity of the lungs | From enrollment to the end of treatment at 4 to 6 weeks
  Diffusing capacity is a measure of how well oxygen and carbon dioxide are transferred (diffused) between the lungs and the blood, and can be a useful test in the diagnosis and to monitor treatment of lung diseases.
Quality of life as measured by the SF-36 questionnaire | On enrollment, after 3 and 6 months from the end of rehabilitation program
  The 36-Item Short Form Survey (SF-36) is an outcome measure instrument that is often used, well-researched, self-reported measure of health. It stems from a study called the Medical Outcomes Study for the objective measure of the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Oksana Kamenskaya, PhD, MD, Principal Investigator — Meshalkin National Research Center
Locations (1):
- Meshalkin Scientific Research Center of the Ministry of Health of Russia, Novosibirsk, Novosibirsk Oblast, Russia